CLINICAL TRIAL: NCT06573710
Title: Correlation Between Postoperative Pain and Apical Extrusion of Different Irrigation Activation Techniques (Randomized Controlled Trial - an In Vitro Study)
Brief Title: Correlation Between Postoperative Pain and Apical Extrusion of Different Irrigation Activation Techniques
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AinShams Uni Endodontics
Record Dates: First submitted 2024-08-24; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Pulpitis - Irreversible
Keywords: irrigant , ultrasonic, LASER , sonic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sonic activation (Experimental)
  Interventions: Device: sonic activator
- LASER activation (Experimental)
  Interventions: Device: LASER activation
- Ultrasonic activation (Experimental)
  Interventions: Device: Ultrasonic activation
- passive irrigation with Endodontic needle (Active Comparator)
  Interventions: Device: passive irrigation with Endodontic needle

INTERVENTIONS:
Device: sonic activator — Polyamide EDDY tips 28mm long is inserted in the canal 2mm short of the working length operated at 6,000 Hz. Activation is done for three cycles each for 20sec. The tip is moved vertically in up and down motion, 1ml is used for each activation cycle followed by 2ml 17% EDTA20
  Arms: Sonic activation
Device: LASER activation — Diode laser 980nm is used to activate the irrigant using fiber optic tip of (200micrometer) and power of 1.5w continuous mode. The tip is placed 2 mm shorter than the working length. Laser irradiation is done for each canal for 20 secs repeated over three cycles for total time of 60 secs and 10 secs pauses between each cycle
  Arms: LASER activation
Device: Ultrasonic activation — ED60tip is used with ultrasonic device operated on mode E and inserted in the canal 2mm short of the working. Activation is done for three cycles each for 20 sec. The tip is moved vertically in up and down motion,1ml is used for each activation cycle followed by 2ml 17% EDTA
  Arms: Ultrasonic activation
Device: passive irrigation with Endodontic needle — Each canal is irrigated with side vented endodontic needle 30G Placed 2mm short of the working length with total time of 60 secs followed by 2ml 17% EDTA
  Arms: passive irrigation with Endodontic needle

SUMMARY:
The aim of this clinical trial is :

To evaluate effect of different techniques of irrigant activation:

1. LASER activation
2. sonic activation
3. ultrasonic activation
4. passive needle irrigation

On:

1. Postoperative pain in vital teeth (Randomized controlled trial)
2. Amount of apical extrusion (In vitro study) Participants will describe their preoperative pain and postoperative pain level at fixed time interval Research will compare postoperative pain accompanied with different irrigant activation techniques and correlate it to amount of debris extrusion

ELIGIBILITY:
Inclusion Criteria:

* Age group 18-50 years
* Males and females
* Lower molars with symptomatic irreversible pulpitis without apical periodontitis

Exclusion Criteria:

* Patients with uncontrolled health conditions
* Immunocompromised patients
* Teeth with periodontal diseases
* Teeth with calcified canals
* pregnant patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of postoperative pain | 8,24,48 hours and one week
  visual analogue scale

SECONDARY OUTCOMES:
Frequency of analgesic intake | 8,24,48 hours and one week
  number of tablets

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided